CLINICAL TRIAL: NCT00337324
Title: Clinical Assessment of Transcutaneous Neurostimulation and Biofeedback (FREMS)in Patients With Diabetic Neuropathy
Brief Title: Electromagnetic Stimulation (FREMS) in Patients With Painful Diabetic Neuropathy
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: IRCCS San Raffaele (Other)
Collaborators: Lorenz Biotech S.p.A. (Industry); University Of Perugia (Other)
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: LORENZ/01
Record Dates: First submitted 2006-06-14; First posted 2006-06-15 (Estimated); Last update posted 2006-06-15 (Estimated); Status verified 2002-03

CONDITIONS: Painful Diabetic Neuropathy
Keywords: Diabetic neuropathy; Complications of diabetes; Neuropathies; Electromagnetic stimulation; Neuropathic pain
MeSH Terms: conditions — Diabetic Neuropathies; Neuralgia

INTERVENTIONS:
Device: Frequency-modulated electromagnetic neural stimulation

SUMMARY:
We postulate that frequency-modulated electromagnetic stimulation (FREMS) may decrease pain in patients with painful diabetic neuropathy.

DETAILED DESCRIPTION:
The stuy was designed as a randomized, double-blind, placebo-controlled cross-over trial. Each patient received two series of ten treatments of either FREMS or placebo in random sequence, with each series lasting no more than three weeks. Primary outcomes (daytime and night-time pain scores) an secondary outcomes (Motor and sensory nerve conduction velocity, sensory tactile perception, foot vibration perception threshold, quality of life, cutaneous microvascular flow, partial tissue tension of oxygen and carbon dioxide) were measured at baseline, after FREMS/placebo series and after 4 months follow-up.

ELIGIBILITY:
Inclusion Criteria:

* type 1 or type 2 diabetes (American Diabetes Association criteria)
* painful diabetic neuropathy with reduced sensory/motor nerve conduction velocity (i.e., <40 m/sec in at least one nerve trunk of the lower limbs)
* vibration perception at the big toe >25 V

Exclusion Criteria:

* presence of any concomitant severe disease
* pregnancy
* renal disease (serum creatinine >2.0 mg/dL)
* history or current foot ulcer
* lower limb arterial disease (ankle-brachial index <0.9) or transcutaneous partial pressure of oxygen <50 mmHg)

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 38
Dates: Start 2002-03; Study Completion 2004-05

PRIMARY OUTCOMES:
Daytime and night-time pain scores assessed at baseline, after FREMS/placebo, and 4 month follow-up

SECONDARY OUTCOMES:
Measurements of the following parameters were made at baseline, after FREMS/placebo, and 4 month follow-up:
Motor and sensory nerve conduction velocity
Sensory tactile perception by monofilament
Foot vibration perception threshold by biothesiometer
Quality of life by SF-36 instrument
Cutaneous microvascular flow by laser doppler
Partial tissue tension of oxygen and carbon dioxide by oxymetry

CONTACTS AND LOCATIONS:
Overall Officials: Emanuele Bosi, MD, Principal Investigator — San Raffaele Scientific Institute and Vita-Salute San Raffaele University, Milano (Italy)
Locations (1):
- San Raffaele Hospital and Scientific Institute, Milan, (Mi), Italy

REFERENCES:
- [Result] Bosi E, Conti M, Vermigli C, Cazzetta G, Peretti E, Cordoni MC, Galimberti G, Scionti L. Effectiveness of frequency-modulated electromagnetic neural stimulation in the treatment of painful diabetic neuropathy. Diabetologia. 2005 May;48(5):817-23. doi: 10.1007/s00125-005-1734-2. Epub 2005 Apr 15. PMID 15834546
- [Derived] Conti M, Peretti E, Cazzetta G, Galimberti G, Vermigli C, Pola R, Scionti L, Bosi E. Frequency-modulated electromagnetic neural stimulation enhances cutaneous microvascular flow in patients with diabetic neuropathy. J Diabetes Complications. 2009 Jan-Feb;23(1):46-8. doi: 10.1016/j.jdiacomp.2008.02.004. Epub 2008 Apr 10. PMID 18403219